CLINICAL TRIAL: NCT06833996
Title: The Efficacy of Bakuchiol in Treating Post-inflammatory Hyperpigmentation
Brief Title: The Efficacy of Bakuchiol in Treating PIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Senior Staff Physician, Henry Ford Health System
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #9920 Protocol 2
Record Dates: First submitted 2016-09-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Post Inflammatory Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation | interventions — bakuchiol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bakuchiol (Experimental): Bakuchiol cream to be applied to a select acne induced PIH spot and a select TCA induced PIH spot
  Interventions: Drug: Bakuchiol
- Vehicle (Placebo Comparator): Vehicle cream to be applied to a select acne induced PIH spot and a select TCA induced PIH spot
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Bakuchiol — Apply bakuchiol cream twice daily to a select acne induced and TCA induced PIH spot for a total of 28 days
  Arms: Bakuchiol
Drug: Vehicle — Apply vehicle cream twice daily to a select acne induced and TCA induced PIH spot for a total of 28 days
  Arms: Vehicle

SUMMARY:
Post-inflammatory hyperpigmentation (PIH) is an acquired hyper melanosis that occurs after cutaneous inflammation or injury frequently affecting darker skinned individuals. Bakuchiol is derived from plants and has inhibitory effects on melanin synthesis, which makes it a promising therapeutic intervention in the management of PIH. This study aims to evaluate the efficacy of bakuchiol in treating post inflammatory hyperpigmentation using the investigators previously validated model in comparison to acne induced PIH.

DETAILED DESCRIPTION:
Post inflammatory hyperpigmentation (PIH) is an acquired hyper melanosis that occurs after cutaneous inflammation or injury. This process can occur in all skin types but more frequently affects darker skinned patients, such as African Americans, Hispanics, Asians, Native Americans, Pacific Islanders and those of Middle Eastern descent. PIH can occur after infection, allergic reactions, contact dermatitis, some medications, burns, following procedures, or inflammatory disease such as acne. In skin of color, PIH frequently occurs in resolving acne lesions and can persist for months after the acne lesion itself has disappeared. In many cases, the resulting PIH can be more distressing than the original insult.

During the investigators previous study on an in-vivo model for post-inflammatory hyperpigmentation, the investigators investigated the clinical, spectroscopic and histologic characteristics of acne-induced PIH versus irritant induced PIH using Trichloroacetic acid (TCA), 35% solution. From this initial study, the investigators concluded that the similarity of Investigator's Global Assessment scores, and spectroscopic measurements using Diffuse Reflectance Spectroscopy and Colorimetry in both acne and TCA-induced PIH at Day 28 suggest that TCA-induced PIH could be a reproducible model for acne induced PIH.

Bakuchiol is a meroterpene phenol derived from plant sources, such as the leaves and seeds of Psoralea corylifolia and the fruits of Piper longum. It has been reported to have anti-inflammatory, anti-bacterial, and antioxidant properties, as well as cause improvement in photodamaged skin. In-vitro studies on melanin production showed that bakuchiol had inhibitory effects on melanin synthesis, which make it a promising therapeutic intervention in the management of PIH.

This study aims to evaluate the efficacy of bakuchiol in treating post inflammatory hyperpigmentation using the investigators previously validated model in comparison to acne induced PIH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with types IV-VI skin
* Minimum age of 18 years
* Able to understand requirements of the study and risks involved
* Able to sign a consent form.
* Existing facial acne pustules (at least three on the face) with history of post-inflammatory hyperpigmentation

Exclusion Criteria:

* Patients with a recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of PIH judged to be clinically significant by the investigator
* Patients with a history of cystic acne or acne conglobate
* Patients on systemic antibiotics or keratolytics (isotretinoin, etc), or topical antibiotics or keratolytic use (retinoids, benzoyl peroxide) over target areas who are unwilling to stop these medications for the duration of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
The degree of hyperpigmentation after treatment with bakuchiol | 56 days
  Pigment will be determined using an Investigators Global Assessment scale
  IGA Hyperpigmentation Description of Hyperpigmentation 0 Clear of hyperpigmentation
  1. Almost clear of hyperpigmentation
  2. Mild, but noticeable hyperpigmentation
  3. Moderate hyperpigmentation (medium brown in quality)
  4. Severe hyperpigmentation (dark brown in quality)
  5. Very severe hyperpigmentation (very dark brown, almost black in quality)

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 3031 West Grand Boulevard,, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor S, Grimes P, Lim J, Im S, Lui H. Postinflammatory hyperpigmentation. J Cutan Med Surg. 2009 Jul-Aug;13(4):183-91. doi: 10.2310/7750.2009.08077. PMID 19706225
- [Background] Davis EC, Callender VD. Postinflammatory hyperpigmentation: a review of the epidemiology, clinical features, and treatment options in skin of color. J Clin Aesthet Dermatol. 2010 Jul;3(7):20-31. PMID 20725554
- [Background] Baumann L, Rodriguez D, Taylor SC, Wu J. Natural considerations for skin of color. Cutis. 2006 Dec;78(6 Suppl):2-19. PMID 17354519
- [Background] Grimes PE, Stockton T. Pigmentary disorders in blacks. Dermatol Clin. 1988 Apr;6(2):271-81. PMID 3378372
- [Background] Chaudhuri RK, Bojanowski K. Bakuchiol: a retinol-like functional compound revealed by gene expression profiling and clinically proven to have anti-aging effects. Int J Cosmet Sci. 2014 Jun;36(3):221-30. doi: 10.1111/ics.12117. Epub 2014 Mar 6. PMID 24471735
- [Background] Polakova K, Fauger A, Sayag M, Jourdan E. A dermocosmetic containing bakuchiol, Ginkgo biloba extract and mannitol improves the efficacy of adapalene in patients with acne vulgaris: result from a controlled randomized trial. Clin Cosmet Investig Dermatol. 2015 Apr 10;8:187-91. doi: 10.2147/CCID.S81691. eCollection 2015. PMID 25914553
- [Background] Ohno O, Watabe T, Nakamura K, Kawagoshi M, Uotsu N, Chiba T, Yamada M, Yamaguchi K, Yamada K, Miyamoto K, Uemura D. Inhibitory effects of bakuchiol, bavachin, and isobavachalcone isolated from Piper longum on melanin production in B16 mouse melanoma cells. Biosci Biotechnol Biochem. 2010;74(7):1504-6. doi: 10.1271/bbb.100221. Epub 2010 Jul 7. PMID 20622433